CLINICAL TRIAL: NCT02789462
Title: Multicenter LAser VA Registry of Percutaneous Coronary Interventions (LAVA)
Acronym: LAVA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bavana V. Rangan, Faculty Associate, Cardiology Research, North Texas Veterans Healthcare System
Other Study IDs: 15075
Record Dates: First submitted 2016-03-22; First posted 2016-06-03 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Arteriosclerosis; Coronary Artery Disease; Laser-assisted Percutaneous Coronary Interventions
MeSH Terms: conditions — Arteriosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing laser-assisted PCI: Patients of VAMC centers who undergone laser-assisted percutaneous coronary interventions.
  Interventions: Procedure: Laser-assisted percutaneous coronary interventions

INTERVENTIONS:
Procedure: Laser-assisted percutaneous coronary interventions — Chart review and data collection of patients undergoing laser-assisted percutaneous coronary interventions

SUMMARY:
This is a multi-center, investigator initiated study that will prospectively and retrospectively examine treatment strategies and outcomes of patients who underwent percutaneous coronary interventions (PCI).

The goal of this multi-center, investigator initiated, registry is to collect information on treatment strategies and outcomes of consecutive patients undergoing laser-assisted PCI among various participating centers. The study is a purely observational, chart review study and involves retrieval and compiling of data based on clinically indicated procedures and follow-up clinical and procedural outcomes.

The information collected will be used to determine the frequency of laser-assisted PCI performed at the participating sites and examine the procedural strategies utilized, and the procedural (both immediate and subsequent) outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone/will be undergoing laser-assisted PCI at each of the participating centers during the study period.
* Willing and able to provide informed consent.

Exclusion Criteria:

* Not eligible candidate as per review by Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects may or may not be patients of each site investigator and they will have undergone clinically indicated laser-assisted PCI at the investigator's site.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Procedural success of the PCI | through hospital discharge post-PCI procedure, approximately 24 hours, but variable based on patient recovery.
  Procedural success is defined as achievement of technical success with no in-hospital major adverse cardiac events (MACE). In-hospital MACE includes any of the following adverse events prior to hospital discharge: death from any cause, myocardial infarction, urgent repeat target vessel revascularization with PCI or coronary bypass surgery, tamponade requiring pericardiocentesis or surgery, or stroke.

SECONDARY OUTCOMES:
Technical success of the PCI | through end of PCI of procedure, approximately 5 minutes after end of procedure
  Technical success of the PCI was defined as successful revascularization with achievement of <30% residual diameter stenosis within the treated segment and restoration of TIMI grade 3 antegrade flow.
major adverse cardiovascular events | through hospital discharge post-PCI procedure,approximately 24 hours, but variable based on patient recovery.
  In-hospital major adverse cardiovascular events (MACE) include any of the following adverse events prior to hospital discharge: death from any cause, myocardial infarction, urgent repeat target vessel revascularization with PCI or coronary bypass surgery, tamponade requiring pericardiocentesis or surgery, or stroke. MACE during clinical follow-up include death, myocardial infarction, target lesion and target vessel revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Bavana Rangan, BDS, MPH, Principal Investigator — UT Southwestern Medical Center/ Dallas VA Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeroudi OM, Alomar ME, Michael TT, El Sabbagh A, Patel VG, Mogabgab O, Fuh E, Sherbet D, Lo N, Roesle M, Rangan BV, Abdullah SM, Hastings JL, Grodin J, Banerjee S, Brilakis ES. Prevalence and management of coronary chronic total occlusions in a tertiary Veterans Affairs hospital. Catheter Cardiovasc Interv. 2014 Oct 1;84(4):637-43. doi: 10.1002/ccd.25264. Epub 2013 Nov 13. PMID 24142769
- [Background] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Background] Boatman DM, Saeed B, Varghese I, Peters CT, Daye J, Haider A, Roesle M, Banerjee S, Brilakis ES. Prior coronary artery bypass graft surgery patients undergoing diagnostic coronary angiography have multiple uncontrolled coronary artery disease risk factors and high risk for cardiovascular events. Heart Vessels. 2009 Jul;24(4):241-6. doi: 10.1007/s00380-008-1114-1. Epub 2009 Jul 22. PMID 19626394
- [Background] Niccoli G, Belloni F, Cosentino N, Fracassi F, Falcioni E, Roberto M, Panico RA, Mongiardo R, Porto I, Leone AM, Burzotta F, Trani C, Crea F. Case-control registry of excimer laser coronary angioplasty versus distal protection devices in patients with acute coronary syndromes due to saphenous vein graft disease. Am J Cardiol. 2013 Nov 15;112(10):1586-91. doi: 10.1016/j.amjcard.2013.07.015. Epub 2013 Aug 30. PMID 23993124
- [Background] Fernandez JP, Hobson AR, McKenzie D, Shah N, Sinha MK, Wells TA, Levy TM, Swallow RA, Talwar S, O'Kane PD. Beyond the balloon: excimer coronary laser atherectomy used alone or in combination with rotational atherectomy in the treatment of chronic total occlusions, non-crossable and non-expansible coronary lesions. EuroIntervention. 2013 Jun 22;9(2):243-50. doi: 10.4244/EIJV9I2A40. PMID 23454891
- [Background] Badr S, Ben-Dor I, Dvir D, Barbash IM, Kitabata H, Minha S, Pendyala LK, Loh JP, Torguson R, Pichard AD, Waksman R. The state of the excimer laser for coronary intervention in the drug-eluting stent era. Cardiovasc Revasc Med. 2013 Mar-Apr;14(2):93-8. doi: 10.1016/j.carrev.2012.12.008. Epub 2013 Jan 16. PMID 23332778
- [Background] Mauri L, Hsieh WH, Massaro JM, Ho KK, D'Agostino R, Cutlip DE. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med. 2007 Mar 8;356(10):1020-9. doi: 10.1056/NEJMoa067731. Epub 2007 Feb 12. PMID 17296821
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284